CLINICAL TRIAL: NCT04917172
Title: Post-Operative Acute Pancreatitis After Pancreaticoduodenectomy: A Prospective Study in the Setting of a High-volume Center.
Brief Title: Post-Operative Acute Pancreatitis After Pancreaticoduodenectomy
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Other Study IDs: Prog. 2130CESC
Record Dates: First submitted 2020-02-17; First posted 2021-06-08 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2021-05

CONDITIONS: Acute Pancreatitis; Pancreatic Fistula; Postoperative Complications
Keywords: PPAP, POH, pancreatoduodenectomy
MeSH Terms: conditions — Pancreatitis; Pancreatic Fistula; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pancreaticoduodenectomy patients: Patients scheduled to receive elective Pancreaticoduodenectomy (PD) (according to Kausch-Whipple or Longmire-Traverso) for all kinds of pancreatic disease (benign, malignant or premalignant) will be enrolled, after having signed a proper informed consent. Each patient will undergo PD once checked the presence of a resectable mass as provided by the normal clinical practice through high-quality cross-sectional imaging. Pre-operative management will follow institutional standards, serum pancreatic amylase and lipase activity will be measured as a part of the standard pre-operative evaluation.
  Interventions: Diagnostic Test: postoperative acute pancreatitis evaluation

INTERVENTIONS:
Diagnostic Test: postoperative acute pancreatitis evaluation — Surgical resection and reconstruction will be carried out according to the Institutional standards. After the surgical procedure, serum pancreatic amylase and lipase activity will be systematically measured two hours after surgery on postoperative day (POD) 0 and every day at 7 a.m. until POD 5 according to our institutional policy. At our institution, the upper limit of normal for serum pancreatic amylase is 52 U/L and for serum lipase is 60 U/L. Postoperative protocols included the routine measurement of inflammatory markers (white blood cell [WBC] count and C-Reactive Protein [CRP]). A urine trypsinogen strip test will be done on POD 1. A trypsinogen-2 concentration of more than 50 µg/l is considered a positive test. As routine clinical practice, a post-operative imaging will be scheduled to check for potential surgical morbidity. Abdominal magnetic resonance imaging (MRI) will be assessed on POD 3.

SUMMARY:
The occurrence of post-pancreatectomy acute pancreatitis (PPAP) can critically impact outcomes after pancreaticoduodenectomy. Although diagnosing a PPAP can be challenging, its identification appears crucial as it can trigger additional morbidity. However, due to the early onset in the perioperative period, the actual spectrum of its early phases has not been systematically explored yet. For this reason, the present study will compare some early biochemical evidence of pancreatic stump damage to morphological changes evident at postoperative imaging.

The postoperative evaluation of serum and/or urine pancreatic enzymes and the radiologic assessment are included in everyday clinical practice. However, the timing and the clinical relevance of such findings mostly rely on the single-institution experience.

This study aims to characterize PPAP by investigating its early radiologic, biochemical, and clinical spectrum of either local or systemic changes associated.

DETAILED DESCRIPTION:
The occurrence of an acute inflammatory process of the pancreatic parenchyma after pancreatic resections has been reported in the literature, but the actual existence of a clinically evident post-pancreatectomy acute pancreatitis (PPAP), defined as a distinct postoperative complication, has been traditionally challenged or, at least, considered to be a rare event.

Emerging evidence, however, defines PPAP as an acute inflammatory/ischemic condition of the pancreatic remnant, able to trigger further postoperative morbidity.

The assessment of ischemic damage of the organ subjected to surgery was also evaluated in other scenarios, such as for the post-cardiac surgery myocardial infarction (MI) and the post-neurosurgery stroke. These ischemic complications, besides having well-defined biochemical features, maybe detected early on post-operative magnetic resonance imaging (MRI). The decrease of pancreatic perfusion may, in some instances, lead to an altered signal in diffusion-weighted images (DWI) and apparent diffusion coefficient (ADC) maps. DWI MRI with Intravoxel incoherent motion (IVIM) sequences have also recently emerged as a key tool to provide quantitative estimates of physiological parameters associated with perfusion and permeability in vivo and can provide information on alterations of tissue cellularity, membrane-cell integrity, and the extracellular space.

The recent PPAP definition has left some unsolved issues, including the need to investigate the role of lipases as a diagnostic criterion, the actual spectrum of PPAP complications, the proper timing for postoperative radiological evaluation, and the preferred imaging modality for PPAP assessment.

ELIGIBILITY:
Inclusion Criteria:

* Male and females ≥ 18 years;
* Scheduled for elective PD;
* ASA score < 4;
* High-quality preoperative cross-sectional imaging of the abdomen performed roughly within one month before surgery;
* Upfront or after neoadjuvant therapy surgery is allowed;
* Ability of the subject to understand the character and individual consequences of the clinical trial;
* Written informed consent.

Exclusion Criteria:

* Patients undergoing emergency surgery;
* Patients with high serum pancreatic amylase or lipase before surgery;
* Chronic use of steroids;
* Informed consent withdrawal;
* Pancreaticogastrostomy (PG);
* Use of octreotide analogs;
* Inability to perform the resection for any reason;
* Total or distal pancreatectomy;
* Need to extend the resection to the pancreas body for any reason.
* Inability to undergo MRI because of contraindications (e.g. claustrophobia, presence of non-MRI-compatible metal implants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to receive elective PD (only Kausch-Whipple or Longmire-Traverso) for all kinds of pancreatic disease (benign, malignant or premalignant) will be enrolled, after having signed a proper informed consent. Each patient will undergo PD once checked the presence of a resectable mass as provided by the normal clinical practice through high-quality cross-sectional imaging. Pre-operative management will follow institutional standards, serum pancreatic amylase and lipase activity will be measured as a part of the standard pre-operative evaluation.
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
the difference in apparent diffusion coefficient (ADC) values at diffusion-weighted (DW) MRI in the PPAP group compared to patients without PPAP. | postoperative day 3 (72 h after the index surgery).
  DW-MRI studies will be performed on a 1.5 T scanner using a multi-channel phased-array torso coil.

SECONDARY OUTCOMES:
intraindividual correlation between longitudinal assessment of serum pancreatic enzymes | 5 days after surgery
  correlation between repeated measurements of serum pancreatic amylase and lipase activity.
postoperative acute pancreatitis and morbidity | 90 days after surgery
  to assess the correlation between the incidence of postoperative acute pancreatitis and the % of patients with postoperative morbidity (scored with the Clavien Dindo Classification of surgical complications)
Postoperative acute pancreatitis incidence | 90 days after surgery
  PPAP as defined by ISGPS

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Marchegiani, MD, PhD, Study Director — Universita di Verona
Locations (1):
- Verona University Hospital, Verona, VR, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bannone E, Andrianello S, Marchegiani G, Malleo G, Paiella S, Salvia R, Bassi C. Postoperative hyperamylasemia (POH) and acute pancreatitis after pancreatoduodenectomy (POAP): State of the art and systematic review. Surgery. 2021 Feb;169(2):377-387. doi: 10.1016/j.surg.2020.04.062. Epub 2020 Jul 5. PMID 32641279
- [Background] Bannone E, Andrianello S, Marchegiani G, Masini G, Malleo G, Bassi C, Salvia R. Postoperative Acute Pancreatitis Following Pancreaticoduodenectomy: A Determinant of Fistula Potentially Driven by the Intraoperative Fluid Management. Ann Surg. 2018 Nov;268(5):815-822. doi: 10.1097/SLA.0000000000002900. PMID 30004917
- [Background] Partelli S, Tamburrino D, Andreasi V, Mazzocato S, Crippa S, Perretti E, Belfiori G, Marmorale C, Balzano G, Falconi M. Implications of increased serum amylase after pancreaticoduodenectomy: toward a better definition of clinically relevant postoperative acute pancreatitis. HPB (Oxford). 2020 Nov;22(11):1645-1653. doi: 10.1016/j.hpb.2020.03.010. Epub 2020 Apr 11. PMID 32291175
- [Background] Chen H, Wang W, Ying X, Deng X, Peng C, Cheng D, Shen B. Predictive factors for postoperative pancreatitis after pancreaticoduodenectomy: A single-center retrospective analysis of 1465 patients. Pancreatology. 2020 Mar;20(2):211-216. doi: 10.1016/j.pan.2019.11.014. Epub 2019 Nov 27. PMID 31831390
- [Background] Loos M, Strobel O, Dietrich M, Mehrabi A, Ramouz A, Al-Saeedi M, Muller-Stich BP, Diener MK, Schneider M, Berchtold C, Feisst M, Hinz U, Mayer P, Giannakis A, Schneider D, Weigand MA, Buchler MW, Hackert T. Hyperamylasemia and acute pancreatitis after pancreatoduodenectomy: Two different entities. Surgery. 2021 Feb;169(2):369-376. doi: 10.1016/j.surg.2020.07.050. Epub 2020 Sep 25. PMID 32981689